CLINICAL TRIAL: NCT06945835
Title: Can a High Intensity Exercise Program for People With Neurologic Disabilities Run by Doctoral of Physical Therapy Students Improve Mobility in Everyday Life
Brief Title: High Intensity Exercise and Improving Physical Activity Among People With Neurologic Dysfunction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Hartford (Other)
Responsible Party: Principal Investigator, Mary Gannotti, Professor, University of Hartford
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 24-10-371
Record Dates: First submitted 2025-02-18; First posted 2025-04-25 (Actual); Last update posted 2025-11-03 (Actual); Status verified 2025-10

CONDITIONS: Cerebral Palsy (CP); Stroke; Spinal Cord Injury; Traumatic Brain Injury; Charcot Marie Tooth Disease (CMT); Spina Bifida
Keywords: high intensity exercise; physical activity; physical disability
MeSH Terms: conditions — Cerebral Palsy; Stroke; Spinal Cord Injuries; Brain Injuries, Traumatic; Charcot-Marie-Tooth Disease; Spinal Dysraphism; Motor Activity

STUDY DESIGN:
Intervention Model Description: Pre test post test design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention Arm (Experimental): Participants will receive two times a week for 8 weeks one hour of individualized exercise program that is based on clinical practice guidelines for high intensity exercise.
  Interventions: Behavioral: Participate in high intensity exercise of at least 20 minutes in 60 minutes session of RPE greater than 6.

INTERVENTIONS:
Behavioral: Participate in high intensity exercise of at least 20 minutes in 60 minutes session of RPE greater than 6. — Partticipants will be performing supported and unsupported walking, free weights, rowing, cycling, resistance bands, adaptive bikes and body weight exercises.

SUMMARY:
The Hawks in Motion (HIM) High Intensity Exercise program is designed to implement the American Physical Therapy Clinical Practice Guidelines and American College of Sports Medicine recommendations for exercise for people with neurologic disability. Doctor of Physical Therapy (DPT) students administer the HIM High Intensity Exercise Program. A prior study evaluated the feasibility, safety, and efficacy of the HIM High Intensity Exercise Program and found it feasible, safe, and effective for 30 people with neurologic disabilities between the ages of 8-99 years. The investigators would like to evaluate whether participation in the HIM High Intensity Exercise Program affects mobility in everyday life. Physical activity will be measured one week before program implementation and one week after to assess if the participants' mobility in everyday improved.

DETAILED DESCRIPTION:
The neurological conditions of spinal cord injury (SCI), stroke (CVA), traumatic brain injury (TBI), cerebral palsy (CP), Charcot-Marie-Tooth (CMT), and Parkinson's disease (PD) create a variety of physical impairments that make movement difficult. For example, people with SCI can have complete or partial paralysis of the arms, legs, and or trunk depending on the location and severity of injury. People with CMT have paralysis in specific muscles of the hands, feet, and trunk. Similarly, people with TBI, CVA, and CP can experience increased muscle tone, decreased voluntary movement, and difficulty moving at correct speeds. This makes walking, moving surface to surface, and doing other physical activities difficult, frustrating, and tiring. People tend not to move, and end up with chronic pain, heart disease, diabetes, and poor health. Physical inactivity is one of the most concerning issues among individuals with chronic neurological conditions, often resulting in limited community participation and reduced quality of life. Many individuals with these conditions struggle to achieve sufficient physical activity levels necessary for functional independence and movement in the community, essential for maintaining social connections and overall well-being. Despite the known benefits of moderate-to-vigorous physical activity, challenges persist in improving mobility in community settings. It has been hypothesized that by increasing function and endurance, which the HIM High Intensity Program can do, mobility in everyday life may improve. The purpose of the project is to see if physical activity among individuals with chronic neurological disabilities can be increased by participation in a community-based exercise program. The investigators would like to answer the following research question: Does participation in an 8-week, twice-a-week high-intensity exercise program for people with neurologic disability run by Doctor of Physical Therapy students increase physical activity in the everyday life?

ELIGIBILITY:
Inclusion Criteria:

* physical disability that limits mobility and activities of daily living, and a neurodevelopmental disability OR neurological disability,
* age 8-99 years of age,
* understands verbal instructions,
* able to obtain medical clearance,
* able to obtain transportation to campus,
* have a parent/guardian/caregiver on site if not own legal authorized representative,
* English speaking.

Exclusion Criteria:

* no presence of a physical disability that impacts activities of daily living, no neurodevelopmental or neurological disability as an underlying cause,
* no person-centered goals (locomotion, fitness, transfers, and mobility),
* unstable cardiac condition,
* uncontrolled seizures,
* unstable oxygen saturation levels,
* no clearance from primary care physician for exercise,
* unable to read and understand English,
* pursuing active litigation for their physical condition.

Ages: 8 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2025-02-24 (Actual); Primary Completion 2025-05-27 (Actual); Study Completion 2025-05-27 (Actual)

PRIMARY OUTCOMES:
Functional Gait Assessment-(FGA) | Baseline and through study completion, an average of 8 weeks
  The Functional Gait Assessment assesses postural stability during walking and assesses an individual's ability to perform multiple motor tasks while walking, with rating of performance on a scale of 0-30, with higher scores indicating better performance. The tool is reliable and valid and has an established minimally clinical important difference (MCID) for the included diagnoses: stroke, vestibular disorders, older adults and geriatric care, Parkinson's Disease, and other non-specific patient populations. For those who cannot complete this test, they will do the Berg Balance Test.
Canadian Occupational Performance Measure (COPM) | Baseline and through study completion, an average of 8 weeks
  The Canadian Occupational Performance Measure is a semi-structured Interview by which participants rate satisfaction and performance on patient-identified goals a scale of 1 to 10, with 1 being the lowest and 10 being the highest.
Berg Balance Scale- (BBS) | Baseline and through study completion, an average of 8 weeks
  The Berg Balance Scale evaluates one's ability to maintain a position and perform a specific task. The scale for scoring is based on a 5-point scale 0 being unable to complete 4 being able to complete, scores ranging 0-70. Higher scores indicate better performance. There are 14 items on the test including; sitting to standing, standing unsupported, sitting with back unsupported, standing to sitting, transfers, standing unsupported with eyes closed, standing unsupported feet together, reaching forward with outstretched arm while standing, pick up object from floor from standing, turning to look behind over both shoulders, 360 turn, toe touch unsupported, tandem unsupported, and single leg stance. The tool is reliable and valid and has an established MCID for the included diagnoses: stroke, SCI, and Parkinson's patients.
Activities-Specific Balance Confidence Scale (ABS) | Baseline and through study completion, an average of 8 weeks
  The Activities Balance Scale is a self-report measure of balance confidence in performing various activities without losing balance or experiencing a sense of unsteadiness, with 16 items. Each item is rated from 0% to 100%, with 0 indicating no confidence and 100% indicating complete confidence. All items are averaged for a total balance confidence score of 0-100%. Higher scores overall indicate greater balance confidence.
10 Meter Walk Test- (10MWT) | Baseline and through study completion, an average of 8 weeks
  The 10-meter walk test is a clinical assessment used to measure short-duration walking speed in meter per seconds (m/s). It involves measuring the time it takes a participant to walk 10 meters, often with a focus on the middle 6 meters to minimize the effects of acceleration and deceleration. Average gait speed is 1.2 m/s, and can be as low as 0.3 in populations with an assistive device. A faster gait speed, or a score of less time indicates better performance. The test is frequently used to assess gait speed in various populations, including those with conditions like stroke, Parkinson's disease, and dementia.
5 Times Sit to Stand: (5XSTS) | Baseline and through study completion, an average of 8 weeks
  The five time sit to stand aids in quantifying functional lower extremity strength and assessing the participant's movement strategies in performing transitional movements. The participant is instructed to sit up and down five times without using their arms as fast as they can after the clinician says "Go", and the timer stops after the patient sits down for the fifth repetition. Time varies by age group, but scores above 12 seconds may indicate fall risk. A faster speed indicates better performance. This outcome measure can be used within a variety of populations, including vestibular disorders, stroke, Parkinson's Disease, Older Adults, Multiple Sclerosis, Cerebral Palsy, and other non-specific patient populations as well. It has excellent validity and reliability, and the MCID has been established.
Timed 30 second repetition arm curl. | Baseline and through study completion, an average of 8 weeks
  For Individuals who are wheelchair users, and are therefore unable to stand, or who cannot safely perform standing tests a timed arm curl test will be performed. The purpose of this test is to assess upper extremity strength and endurance. The test is conducted using the dominant arm. The participant is seated on a chair with feet flat on the floor, holding a 5-pound weight in a suitcase grip (palm is facing the body) in a vertically down position by the chair (start position). The participant performs an arm curl throughout a full range of motion, gradually turning the palm up and the elbow fully bent. The arm is lowered again to the starting position with the elbow fully straightened. The participant performs as many as possible in 30 seconds. Range of number of arm cults can be from 0-30. The average number varies by age and gender, but a high number repetitions performed in 30 seconds indicates better muscle performance.
Timed 30 second Wheelchair Push Ups. | Baseline and through study completion, an average of 8 weeks
  Participants who use a wheelchair as primary means of locomotion will do timed 30 second wheelchair pushups. The participant demonstrates how many wheelchair pushups can be completed in 30 seconds. A push-up is when the bottom is unweighted from the seat. Range of pushup can be from 0-30. A high number repetitions performed in 30 seconds indicates better muscle performance.
Six minute walk test (6MWT)/6 minute push test) | Baseline and through study completion, an average of 8 weeks
  The 6MWT/push test is a sub-maximal exercise test used to assess walking or locomotion endurance and aerobic capacity. Participants will walk/push a set circuit for a total of six minutes. Distance is measured during the 6MWT or push test. Distances walked can range from 0 to 2500 meters. Longer distances indicate increased endurance and aerobic capacity.

SECONDARY OUTCOMES:
Physical Activity Monitoring | Baseline and through study completion, an average of 8 weeks
  The Actigraph GTX will be used to measure physical activity across 7 days before and after the activity. It will be worn on the waist for people who ambulate and on the wrist for those who use a wheelchair. We will classify the movement patterns into sedentary and moderate to vigorous activity using the software with the accelerometers, and this will be compared pre- and post-intervention. The investigators evaluate average steps, percentage of time in sedentary, light, moderate, vigorous, and very vigorous activity per week. Range of average steps is 0-unlimited and average time spent in sedentary light, moderate, vigorous, and very vigorous activity per week is 0-100% . A higher number of steps with less time in sedentary activity time indicate greater physical activity.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Hartford, West Hartford, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No
none at this time